CLINICAL TRIAL: NCT05392400
Title: The Use of Steri3X for Prevention of Post-operative Wound Infections in Cesarean Sections
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-08663-FB
Record Dates: First submitted 2022-05-22; First posted 2022-05-26 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2022-05

CONDITIONS: Surgical Site Infection; Cesarean Section; Complications, Wound, Infection (Following Delivery); Postpartum Complication
Keywords: Intrauterine infection, cesarean, postpartum endometritis, surgical site infection, postoperative wound infection
MeSH Terms: conditions — Surgical Wound Infection; Wounds and Injuries; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control (Active Comparator): Currently, the standard of care for Cesarean section patients includes covering the closed incision with a sterile bandage to reduce the chance of infection, and approximately 48 hours of post-op hospitalization and wound surveillance. The "control" group will receive post-operative wound dressings consistent with the current standard of care.
  Interventions: Other: Control
- Experimental (Experimental): Patients randomized to the Experimental group will receive treatment with Steri3x immediately following closure of the Cesarean section incision. Participants in the experimental group will receive approximately 48 hours of post-op hospitalization and wound surveillance.
  Interventions: Device: Steri3X

INTERVENTIONS:
Device: Steri3X — This study will initially attempt to recruit pregnant patients at the Regional One Health outpatient obstetrics clinic, at which point they will be randomly assigned to one of two cohorts. Participants who are consented to participate in the study will receive a chart flag in the EMR so that they may receive the proper intraoperative and postoperative treatment(s). Patients randomized to receive the Steri3X wound dressing will have the liquid polymer applied in the operating room after closure of the Cesarean section incision. Participants of both arms will be monitored postoperatively to assess for signs and symptoms of postoperative surgical site infection(s).
  Arms: Experimental
Other: Control — Device: Steri3X
  This study will initially attempt to recruit pregnant patients at the Regional One Health outpatient obstetrics clinic, at which point they will be randomly assigned to one of two cohorts. Participants who are consented to participate in the study will receive a chart flag in the EMR so that they may receive the proper intraoperative and postoperative treatment(s). Patients randomized to receive the control wound dressing will have the current standard of care dressing applied in the operating room after closure of the Cesarean section incision. Participants of both arms will be monitored postoperatively to assess for signs and symptoms of postoperative surgical site infection(s).
  Arms: Control

SUMMARY:
Postpartum infection if a major cause of maternal morbidity and mortality and surgical site infections are some of the common complications following cesarean section. This study aims to determine the effect of Steri3X on the incidence of cesarean section SSI at Regional One Hospital.

DETAILED DESCRIPTION:
Postpartum infection is a major cause of maternal morbidity and prolonged hospitalization, and places a large burden on the healthcare system with an additional cost of $3,700 (Olsen et al., 2010). Surgical site infection (SSI) is one of the most common post-operative complications following cesarean section, with an incidence of 3-15% worldwide (Zuarez-Eaaston et al., 2017). Wound dressings that are applied after closure of a surgical incision may help healing by providing physical support, protection from external contaminants, and by absorbing exudate (Dumville et al., 2016). A new FDA-approved microbicidial liquid adhesive, Steri3X, has been shown to reduce the incidence of pin-tract infection by 100% in a randomized-controlled trial following external fixation in patients undergoing reconstructive surgery for deformity correction (Pema, 2020). Steri3X is reported to be effective against S. aureus (both MSSA and MRSA), Candida albicans, E. coli, P. aeruginosa, and Candida auris, which are common organisms involved in dermatological infections. The most common organisms responsible for cesarean section SSI include enteric gram negative bacilli, enterococci, and group B streptococcus (Gur et al., 2015). The advantage of this polymer following C-sections is unknown, and a larger study is needed to provide a more robust analysis. This study aims to determine the effect of Steri3X on the incidence of cesarean section SSI at Regional One Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 years old or older
* C-section patients only (primary, repeat, or stat)
* Diabetes, obesity ok to include (but not required)
* Patients receiving PCN for GBS prophylaxis ok to include (but not required)
* Application of Steri3X immediately post-op

Exclusion Criteria:

* Chorioamnionitis or other existing infection excluded (Single maternal fever >39 C, 2 maternal fevers > 38, or clinical risk factors for chorioamnionitis)
* Patients receiving antibiotic treatment for existing or prior infection other than PCN for GBS prophylaxis
* Patients receiving Prevena or other wound vac
* Rupture of membranes >24 hours

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-02-07 (Estimated); Primary Completion 2024-02-07 (Estimated); Study Completion 2024-02-07 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection | 8 weeks
  Postoperative patients will be monitored for signs/symptoms of infection after Cesarean section during their inpatient postoperative stay and also during postpartum office visits.

CONTACTS AND LOCATIONS:
Overall Officials: Ramona Phinehas, MD, Study Director — University of Tennessee
Locations (1):
- Regional One Health Medical Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsiung SH, Robins P. Evaluation of a flexible new liquid polymer wound dressing. J Drugs Dermatol. 2005 Sep-Oct;4(5):580-2. PMID 16167416
- [Background] Robins P, Goldberg L, Moy R, Nouri K, Perez M, Saini R, Sarnoff D, Spencer J. The effectiveness of liquid bandage as an adhesive and antimicrobial agent. J Drugs Dermatol. 2008 Aug;7(8):764-6. No abstract available. PMID 18720693
- [Background] Olsen MA, Butler AM, Willers DM, Gross GA, Hamilton BH, Fraser VJ. Attributable costs of surgical site infection and endometritis after low transverse cesarean delivery. Infect Control Hosp Epidemiol. 2010 Mar;31(3):276-82. doi: 10.1086/650755. PMID 20102279
- [Background] Zuarez-Easton S, Zafran N, Garmi G, Salim R. Postcesarean wound infection: prevalence, impact, prevention, and management challenges. Int J Womens Health. 2017 Feb 17;9:81-88. doi: 10.2147/IJWH.S98876. eCollection 2017. PMID 28255256
- [Background] Dumville JC, Gray TA, Walter CJ, Sharp CA, Page T, Macefield R, Blencowe N, Milne TK, Reeves BC, Blazeby J. Dressings for the prevention of surgical site infection. Cochrane Database Syst Rev. 2016 Dec 20;12(12):CD003091. doi: 10.1002/14651858.CD003091.pub4. PMID 27996083
- See also: Shital Pema, DPM. An Evaluation of the Use of a Novel Microbicidal Liquid Polymer for the Reduction of Pin-tract Infection in Research Participants Receiving External Fixation Following Deformity Correction and Traumatic Provisional Fixation. — https://oatext.com/an-evaluation-of-the-use-of-a-novel-microbicidal-liquid-polymer-for-the-reduction-of-pin-tract-infection-in-external-fixation-procedures-for-deformity-correction.php